CLINICAL TRIAL: NCT00078624
Title: Knee Stability Training in Individuals With Knee Osteoarthritis
Brief Title: Knee Stability Training for Knee Osteoarthritis (OA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIAMS-117; R01AR048760-01A2 (NIH)
Record Dates: First submitted 2004-03-03; First posted 2004-03-04 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Osteoarthritis; Joint Diseases
Keywords: Osteoarthritis; Knee Joint; Joint Stability; Motor Control; Exercise Therapy
MeSH Terms: conditions — Osteoarthritis; Joint Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Traditional exercise program supplemented with knee stability training activities
  Interventions: Other: Knee stability training
- 2 (Active Comparator): Traditional exercise program
  Interventions: Other: Traditional exercise therapy for knee osteoarthritis

INTERVENTIONS:
Other: Traditional exercise therapy for knee osteoarthritis — Exercises include stretching, strengthening, and aerobic exercise
  Arms: 2
Other: Knee stability training — The addition of agility and perturbation training techniques to the traditional exercise program
  Arms: 1

SUMMARY:
People with knee osteoarthritis (OA) frequently complain of knee instability. This study will test whether certain exercises can improve knee stability, reduce pain, and improve physical function in people with knee OA.

Study hypotheses: 1) Participants in the stability training group will demonstrate less pain and higher levels of physical function, based on self-report measures of pain and function (WOMAC, Lower Extremity Function Scale), and less time to complete the Get Up and Go test, a physical performance measure of function. 2) During walking and the step down task, participants in the stability training group will demonstrate greater knee motion during weight bearing, greater vertical ground reaction forces and loading rates, and reduced ratios of co-contraction between quadriceps/hamsting and tibialis anterior/gastrocnemius muscle pairs compared to the standard group. Participants in the stability group will also demonstrate greater step lengths, single limb support times, and average walking velocity compared to the standard group.

DETAILED DESCRIPTION:
Traditional exercise therapy for knee OA primarily focuses on lower limb strength and joint motion deficits. Recent evidence has suggested that changes in lower limb biomechanical factors during weight bearing activities may have substantial impact on physical function and disease progression in individuals with knee OA. The effectiveness of exercise therapy programs might be improved by incorporating balance and agility training techniques (knee stability training). The aim of this trial is to test the effectiveness of supplementing traditional exercise therapy with knee stability training techniques tailored for individuals with knee OA.

Participants will be randomly assigned to one of two groups. The first group will participate in a standard rehabilitation program of traditional exercise therapy for knee OA. The second group will participate in a standard rehabilitation program supplemented with a knee stability program. Study visits will occur at study entry, 2 months, 6 months, and 1 year. At each study visit, changes in pain, physical function, and biomechanical factors will be assessed. This study will last for one year.

ELIGIBILITY:
Inclusion Criteria:

* Meet the 1986 American College of Rheumatology (ACR) clinical criteria for knee osteoarthritis
* Grade II or greater Kellgren and Lawrence radiographic changes

Exclusion Criteria:

* History of two or more falls within the year prior to study entry
* Unable to walk a distance of 100 feet without an assistive device or a rest period
* Total knee arthroplasty
* Uncontrolled hypertension
* History of cardiovascular disease
* History of neurological disorders that affect lower extremity function such as stroke or peripheral neuropathy
* Corticosteroid injection to the quadriceps or patellar tendon in the past month, or 3 or more within the past year
* Quadriceps tendon rupture, patellar tendon rupture, or patellar fracture that could place them at risk of re-injury during quadriceps strength testing
* Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2004-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster OA index (WOMAC) | Measured at baseline, 2 months, 6 months, 1 year
Lower Extremity Function Scale | Measured at baseline, 2 months, 6 months, 1 year
Get Up and Go test (a physical performance measure of function) | Measured at baseline, 2 months, 6 months
Knee Outcome Survey - Activities of Daily Living Scale | Measured at baseline, 2 months, 6 months, 1 year

SECONDARY OUTCOMES:
Cartilage morphology changes as measured by MRI | Measured at baseline, 1 year
Physical Activity Scale for the Elderly | Measured at baseline, 2 months, 6 months, 1 year
Quadriceps strength and activation | Measured at baseline, 2 months, 6 months
Radiographic severity of OA | Measured at baseline, 1 year
Fear Avoidance questionnaire for the knee | Measured at baseline, 2months, 6 months, 1 year
Beck Anxiety Index | Measured at baseline, 2 months, 6 months, 1 year
Center for Epidemiological Studies Depression Scale | Measured at baseline, 2 months, 6 months, 1 year
Motion analysis variables (knee motion, vertical ground reaction force, loading rates, knee adduction/abduction moment, and lower extremity muscle co-contractions during walking and a step-down task) | Measured at baseline, 2 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: G. Kelley Fitzgerald, PhD, PT, Principal Investigator — University of Pittsburgh, Department of Physical Therapy, School of Health and Rehabilitation Sciences
Locations (1):
- University of Pittsburgh, Department of Physical Therapy, School of Health and Rehabilitation Sciences, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Fitzgerald GK, White DK, Piva SR. Associations for change in physical and psychological factors and treatment response following exercise in knee osteoarthritis: an exploratory study. Arthritis Care Res (Hoboken). 2012 Nov;64(11):1673-80. doi: 10.1002/acr.21751. PMID 22674892
- [Derived] Teixeira PE, Piva SR, Fitzgerald GK. Effects of impairment-based exercise on performance of specific self-reported functional tasks in individuals with knee osteoarthritis. Phys Ther. 2011 Dec;91(12):1752-65. doi: 10.2522/ptj.20100269. Epub 2011 Oct 14. PMID 22003157
- [Derived] Fitzgerald GK, Piva SR, Gil AB, Wisniewski SR, Oddis CV, Irrgang JJ. Agility and perturbation training techniques in exercise therapy for reducing pain and improving function in people with knee osteoarthritis: a randomized clinical trial. Phys Ther. 2011 Apr;91(4):452-69. doi: 10.2522/ptj.20100188. Epub 2011 Feb 17. PMID 21330451